CLINICAL TRIAL: NCT04154748
Title: Argon Plasma Coagulation for Barrett's Esophagus With Low Grade Dysplasia: A Randomized Trial With Long Term Follow-up Evaluating the Impact of Power Setting and Proton Pump Inhibitor Dose
Brief Title: Argon Plasma Coagulation for Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0102
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Barretts Esophagus With Low Grade Dysplasia
Keywords: Barretts Esophagus; Dysplasia; Argon Plasma Coagulation; Endoscopic Treatment
MeSH Terms: conditions — Barrett Esophagus | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: Investigator initiated, single-center, parallel-group RCT conducted in a tertiary referral center in Poland.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were blinded to the power settings used for APC, but they knew the PPI dose they received. The endoscopist performing APC ablation was blinded to participant allocation and APC power setting (the power was set up by an assistant who knew the group allocation and the power display remained covered during the entire procedure). The endoscopist and pathologist involved in efficacy assessment were blinded to participant allocation.
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- APC 90W / PPI 120mg (Experimental): treatment with high-power argon plasma coagulation (90 Watt) followed by acid suppression with high-dose oral omeprazole (40 mg t.i.d)
  Interventions: Device: Argon Plasma Coagulation 90W power; Drug: Omeprazole 120 mg
- APC 90W / PPI 40mg (Active Comparator): treatment with high-power argon plasma coagulation (90 Watt) followed by acid suppression with standard dose oral omeprazole (40 mg q.d)
  Interventions: Device: Argon Plasma Coagulation 90W power; Drug: Omeprazole 40 mg
- APC 60 W/ PPI 120mg (Active Comparator): treatment with standard-power argon plasma coagulation (60 Watt) followed by acid suppression with high-dose oral omeprazole (40 mg t.i.d)
  Interventions: Device: Argon Plasma Coagulation 60W power; Drug: Omeprazole 120 mg

INTERVENTIONS:
Device: Argon Plasma Coagulation 90W power
  Arms: APC 90W / PPI 120mg; APC 90W / PPI 40mg
Device: Argon Plasma Coagulation 60W power
  Arms: APC 60 W/ PPI 120mg
Drug: Omeprazole 120 mg
  Arms: APC 60 W/ PPI 120mg; APC 90W / PPI 120mg
Drug: Omeprazole 40 mg
  Arms: APC 90W / PPI 40mg

SUMMARY:
Background and study aims. To evaluate the impact of power setting and proton pump inhibitor (PPI) dose on the efficacy and safety of argon plasma coagulation (APC) of Barrett's esophagus (BE) with low-grade dysplasia (LGD).

Patients and methods. Investigator initiated, single-center, parallel-group randomized controlled trial (RCT) conducted in a tertiary referral center in Poland. Consecutive patients with BE and LGD were randomly assigned to APC with power set at 90 Watt (90W) or 60 Watt (60W) followed by 120 mg or 40 mg omeprazole for six weeks. The primary outcome of the study was the rate of complete (endoscopic and histologic) ablation of BE at six weeks. Secondary outcomes included safety and long-term efficacy (at two years and at the end of a long-term follow-up of over 4 years.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult patients with low-grade dysplasia in flat Barrett's mucosa referred for endoscopic treatment,
* signed an informed consent to participate in the study.

Exclusion Criteria:

* high-grade dysplasia or adenocarcinoma,
* visible lesions (nodules, ulcerations) in Barrett's mucosa,
* serious comorbidities and short life expectancy,
* coagulopathy,
* pregnancy or lactation,
* psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2002-06-04 (Actual); Primary Completion 2015-02-10 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Complete ablation rate 6 weeks after APC treatment. | 6 weeks
  Complete ablation was defined as no endoscopic and histologic evidence of Barrett's mucosa, dysplasia, and buried metaplastic glands

SECONDARY OUTCOMES:
Adverse event rate during APC treatment and within 6-week post-treatment period | 6 weeks
Complete ablation rate two years after APC treatment | 2 years
  Complete ablation was defined as no endoscopic and histologic evidence of Barrett's mucosa, dysplasia, and buried metaplastic glands
Complete ablation rate at the end of follow-up | Long term follow-up (>4 yars)
  Complete ablation was defined as no endoscopic and histologic evidence of Barrett's mucosa, dysplasia, and buried metaplastic glands

REFERENCES:
- [Derived] Wronska E, Polkowski M, Orlowska J, Mroz A, Wieszczy P, Regula J. Argon plasma coagulation for Barrett's esophagus with low-grade dysplasia: a randomized trial with long-term follow-up on the impact of power setting and proton pump inhibitor dose. Endoscopy. 2021 Feb;53(2):123-132. doi: 10.1055/a-1203-5930. Epub 2020 Jul 10. PMID 32650347